CLINICAL TRIAL: NCT01503749
Title: The Role of Peripheral Mononuclear Cells for Treatment of Advanced Liver Cirrhosis
Brief Title: Safety and Efficacy Study of Peripheral Blood Mononucleated Cells for Treatment of Liver Cirrhosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: PBMC
Record Dates: First submitted 2012-01-02; First posted 2012-01-04 (Estimated); Results first posted 2014-12-19 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-10

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Filgrastim; Leukapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Three patients with liver cirrhosis of this arm will not receive any intervention regarding to peripheral blood mononucleated cells.
- G-colony stimulating factor (Active Comparator): G-colony stimulating factor (5ug/kg/day)will be administered twice subcutaneously for 3 days to three patients with liver cirrhosis of this arm.
  Interventions: Drug: G-colony stimulating factor
- Infusion of the mobilized monocyte cells (Experimental): G-colony stimulating factor (5ug/kg/day)will be administered twice subcutaneously for 3 days to three patients with liver cirrhosis of this arm. On the day 4th, leukapheresis will be done to collect peripheral blood mononucleated cells
  . And then we are going to infuse the collected peripheral blood mononucleated cells of their own through the portal vein of each patients under ultrasonographic guidance.
  Interventions: Other: Infusion of the mobilized monocyte cells

INTERVENTIONS:
Drug: G-colony stimulating factor — G-colony stimulating factor (5ug/kg/day)will be administered subcutaneously to three patients with liver cirrhosis of this arm.
  Other Names: Filgrastim
  Arms: G-colony stimulating factor
Other: Infusion of the mobilized monocyte cells — G-colony stimulating factor (5ug/kg/day)will be administered twice subcutaneously for 3 days to three patients with liver cirrhosis of this arm. On the day 4th, leukapheresis will be done to collect peripheral blood mononucleated cells. And then we are going to infuse the collected peripheral blood mononucleated cells of their own through the portal vein of each patients under ultrasonographic guidance.
  Other Names: Filgrastim; leukapheresis
  Arms: Infusion of the mobilized monocyte cells

SUMMARY:
The investigators aim to investigate the safety and efficacy of peripheral blood monocyte for the treatment of patients with advanced liver cirrhosis.

DETAILED DESCRIPTION:
G-colony stimulating factor(5ug/kg/day)will be administered twice subcutaneously for 3 days to three patients with liver cirrhosis. On the day 4th, plasmapheresis will be done to collect peripheral blood mononucleated cells

. And then we are going to infuse the collected peripheral blood mononucleated cells of their own through the portal vein of each patients under ultrasonographic guidance.

ELIGIBILITY:
Inclusion Criteria:

1. 20 =< Age < 80
2. Advanced liver cirrhosis with Child-Pugh score 8 or 9 (including patients who have no radiologic evidence of remnant HCC for more than 2 years after treatment)

Exclusion Criteria:

1. HBsAg-positive
2. Active status of hepatocellular carcinoma (HCC) (except patients who have no radiologic evidence of remnant HCC for more than 2 years after treatment)
3. History of hemochromatosis and/or autoimmune hepatitis
4. Pregnant women or lactating women
5. Hemoglobin < 8g/dL (male), 7.5g/dL (female) or white blood cell (WBC) <1,500 mm3 or Neutrophils <500/mm3 or platelet count <50,000/mm3
6. Serum creatinine> 1.5 x normal upper limit or creatinine clearance <60 ml/min
7. Presence of signs of malignant tumors or tumor suspected symptoms, or history of malignant tumors with recurrence rate greater than 20% within two years
8. Gastrointestinal bleeding within the last 3 months or if there is a history of spontaneous bacterial peritonitis
9. Presence of portal vein thrombosis
10. Presence of acute infections

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-01; Primary Completion 2013-07 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Hwan Yoon, M.D., Ph. D., Principal Investigator — Seoul National University Hospital

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment location: single medical center (Seoul National University Hospital) Recruitment period: between February 2012 and July 2013
Pre-assignment Details: Number of total enrolled pariticipants: 9 Number of screened participants: 14 Number of dropped participants: 5 (Withdraw consent:4, etc:1 due to development of hepatocellular carcinoma) Number of completed participants: 9
Groups:
- Control: Three patients with liver cirrhosis of this arm will not receive any intervention regarding to peripheral blood mononucleated cells
  .
- Infusion of the Mobilized Peripheral Blood Mononucleated Cells: G-colony stimulating factor (5ug/kg/day)will be administered twice subcutaneously for 3 days to three patients with liver cirrhosis of this arm. On the day 4th, leukapheresis will be done to collect peripheral blood mononucleated cells
  . And then we are going to infuse the collected peripheral blood mononucleated cells of their own through the portal vein of each patients under ultrasonographic guidance.
  Infusion of the mobilized peripheral blood mononucleated cells: G-colony stimulating factor (5ug/kg/day)will be administered twice subcutaneously for 3 days to three patients with liver cirrhosis of this arm. On the day 4th, leukapheresis will be done to collect peripheral blood mononucleated cells. And then we are going to infuse the collected peripheral blood mononucleated cells of their own through the portal vein of each patients under ultrasonographic guidance.
Period: Overall Study
Arm/Group | Control | G-colony Stimulating Factor | Infusion of the Mobilized Peripheral Blood Mononucleated Cells
Started | 3 | 3 | 3
Completed | 3 | 3 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | G-colony Stimulating Factor | Infusion of the Mobilized Peripheral Blood Mononucleated Cells | Total
Number analyzed (Participants) | 3 | 3 | 3 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 1 | 5
  >=65 years | 1 | 1 | 2 | 4
Age, Continuous [Mean (Full Range); unit: years] | 57 [45 to 65] | 62 [59 to 68] | 63.3 [54 to 71] | 60.8 [45 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 4
  Male | 2 | 1 | 2 | 5
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 3 | 3 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Severe Adverse Events
Description: No serious adverse event. Minor adverse events (not considered to be related to this study), as follows; Control: 6 events (ascites and pleural tapping, gum bleeding, ascties tapping x3, diarrhea) G-colony stimulating factor group: 6 events (percutaneous vertebroplasty, abdominal pain and nausea, hyperkalemia, ascties tapping, diarrhea, liver transplantation) Infusion of the mobilized peripheral blood mononucleated cells group: 1 event (hepatic encephalopathy)
Time Frame: up to 6 months
Population: Nine patients who fulfilled the inclusion and exclusion criteria.
Measure: Number; unit: participants
Arm/Group | Control | G-colony Stimulating Factor | Infusion of the Mobilized Peripheral Blood Mononucleated Cells
Number analyzed (Participants) | 3 | 3 | 3
participants | 0 | 0 | 0

2. Secondary Outcome: Mean Change in Child-Pugh Score and Model For End-Stage Liver Disease (MELD) Score
Description: The efficacy (mean change in Child-Pugh score and Model For End-Stage Liver Disease score [at weeks 24]) of ultrasound-guided percutaneous portal transplantation of peripheral blood monocyte cell in cirrhotic patients. MELD Score = (0.957 * ln(Serum Cr) + 0.378 * ln(Serum Bilirubin) + 1.120 * ln(INR) + 0.643 ) * 10 (if hemodialysis, value for Creatinine is automatically set to 4.0) (minimum <9: 1.9% mortality; maximum 40 or more: 71.3% mortality). Child-Pugh score = Bilirubin (mg/dl): <2 (1 point),2-3 (2 points), >3 (3 points) + Albumin (g/dl): >3.5 (1 point),3.5-2.8 (2 points), <2.8 (3 points) + PT prolongation (INR): <4 seconds (<1.7) (1 point), 4-6 seconds (1.7-2.3) (2 points),>6 seconds (>2.3) (3 points) + Ascites: Absent (1 point), Slight (2 points), Moderate (3 points) + Encephalopathy: Absent (1 point), Mild (I-II) (2 points), Severe (III-IV) (3 points) ; Class A: 5-6, Class B: 7-9, Class C: 10-15 (minimum 5, maximum 15; higher Child-Pugh score with worse prognosis)
Time Frame: Baseline and Week 24
Population: A total of 9 decompensated cirrhotic patients (5 men and 4 females, age range 45-71 years) grouped by randomization.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Control | G-colony Stimulating Factor | Infusion of the Mobilized Peripheral Blood Mononucleated Cells
Number analyzed (Participants) | 3 | 3 | 3
score
  Baseline Child-Pugh score | 9 (1) | 10 (1) | 9 (1)
  Child-Pugh score at 24 weeks | 9.5 (2.5) | 10 (2) | 8.3 (1.1)
  Baseline MELD score | 15.9 (3.2) | 18.9 (2.2) | 14.4 (2.2)
  MELD score at 24 weeks | 15.5 (3.9) | 24.0 (3.9) | 14.7 (3.4)
Statistical Analysis 1: Comparison: Control vs G-colony Stimulating Factor vs Infusion of the Mobilized Peripheral Blood Mononucleated Cells; Test type: Superiority or Other; p > 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: from the baseline till at week 24
Description: No splenic rupture among the patients who received G-CSF mobilization during the study period (till at week 24).
  No bleeding or infection after portal administration of PBMCs during the study period (till at week 24).
Arm/Group | Control | G-colony Stimulating Factor | Infusion of the Mobilized Peripheral Blood Mononucleated Cells
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 1/3 | 1/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=3) | G-colony Stimulating Factor (N=3) | Infusion of the Mobilized Peripheral Blood Mononucleated Cells (N=3)
hepatic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
ascties tapping (Hepatobiliary disorders) | 2 (4) | 1 (1) | 0 (0)
Liver transplantation (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
hyperkalemia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
percutaneous vertebroplasty (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
gum bleeding (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No